CLINICAL TRIAL: NCT03773003
Title: Pathophysiology of Cancer Related Fatigue (CRF) and Chronic Fatigue (CFS/ME) by Lipidomics, Metabolomics, Microbiome and Exome Analysis and Investigation of Clinical Improvement Under Administration of Probiotics
Brief Title: Research for Pathophysiology of Cancer Related Fatigue (CRF) and Chronic Fatigue (CFS/ME)
Acronym: IMPROFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Principal Investigator, Michael Jelden, Principal Investigator, University Hospital, Saarland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IMPROFA
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cancer Related Fatigue; Fatigue Syndrome, Chronic
Keywords: Cancer Fatigue, Chronic Fatigue
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled intervention with probiotics
  There are three groups in the study:
  1. Tumor disease with fatigue
  2. Tumor disease without fatigue
  3. Healthy control group
Who Masked: Investigator
Masking Description: Blinding will be made at the probiotics manufacturer's establishment. Neither investigators nor care providers nor patients know their status til the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1: Tumor disease w/o fatigue (Active Comparator): Group receiving probiotics.
  Interventions: Dietary Supplement: Probiotics
- Arm 2: Tumor disease w/o fatigue (Placebo Comparator): Group receiving placebo (corn starch)
  Interventions: Dietary Supplement: Placebo
- Arm 3: Healthy control group (Active Comparator): Group receiving probiotics
  Interventions: Dietary Supplement: Probiotics
- Arm 4: Healthy control group (Placebo Comparator): Group receiving placebo (corn starch)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — The administered probiotics are readily available on the market and contain
  * Bifidobacterium breve, B. infantis, B. lactis, B. longum
  * Lactobacillus acidophilus, L. bulgaricus, L. casei, L. crispatus, L. fermentum, L. paracasei, L. plantarum, L. reuteri, L. rhamnosus, L. salivarius
  * Streptococcus thermophilus
  Arms: Arm 1: Tumor disease w/o fatigue; Arm 3: Healthy control group
Dietary Supplement: Placebo — Identically looking to verum, containing corn starch.
  Arms: Arm 2: Tumor disease w/o fatigue; Arm 4: Healthy control group

SUMMARY:
Research for Pathophysiology of Cancer Related Fatigue (CRF) and Chronic Fatigue Syndrome (CFS/ME) by Lipidomics, Metabolomics, Intestinal and Peritoneal Microbiome Analysis and Exome Analysis and Investigation of a Possible Benefit of Probiotics.

DETAILED DESCRIPTION:
This study aims to identify the underlying pathophysiology of Cancer Related Fatigue (CRF) by screening lipidome, metabolome, exome and microbiome of affected patients with tumor disease with and without fatigue. These results will be compared to an age- and gender matched control group with a comparable tumor disease and to another age- and gender matched control group without tumor disease.

The investigators are following the same strategy for investigating an underlying pathophysiology of Chronic Fatigue Syndrome (CFS/ME) in another group of patients. The age- and gender matched control group will be established from the beforementioned control group.

The investigators will also be screening for a peritoneal microbiome (possible correlate for leaky gut) in study patients undergoing abdominal surgery.

We will also investigate changes in fatigue and in lipidome, metabolome, exome and microbiome by double-blinded, placebo-controlled administration of probiotics to the study population.

ELIGIBILITY:
Inclusion Criteria:

* histologically, cytologically or radiologically confirmed tumor disease
* indication for chemotherapy
* Written consent to participation

Exclusion Criteria:

* chronic-inflammatory bowel disease
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of fatigue symptoms | 3 months after end of chemotherapy
  Improvement of fatigue as measured by validated psychometric questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jelden, MD, Principal Investigator — University Hospital, Saarland
Locations (1):
- Saarland University Medical Center, Homburg, Saarland, Germany